CLINICAL TRIAL: NCT04188431
Title: Dexamethasone and Postoperative Bleeding Following Tonsillectomy in Children: Double-blind, Randomized, Placebo Control, Multi-centre, International, Pragmatic, Non-inferiority Trial
Brief Title: Dexamethasone and Postoperative Bleeding Following Tonsillectomy in Children
Acronym: Blueberry
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of finance
Sponsor: Walid HABRE (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Walid HABRE, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2019-02268
Record Dates: First submitted 2019-12-01; First posted 2019-12-05 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pain, Postoperative; Tonsillar Bleeding; Postoperative Nausea and Vomiting
Keywords: reintervention; children
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blind (investigator-surgeon-patient blinded), randomized, placebo control, multi-centre, international, pragmatic, Non-inferiority trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients are allocated by block randomisation using sealed envelope system. An external person dedicated by Sponsor is in charge to randomize groups of treatment allocation through a website-generated list and to conceal the lists. Each centre receives the sealed opaque envelopes which contain treatment allocation. The envelope will be opened just before surgery.
  A member of the team not involved in the anaesthesia care will open an envelope and prepare the tested medication according to the result of randomization (Dexamethasone or NaCl). The repartition ratio between the 2 arms is 1:1 with a block size of 10.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Single intraoperative administration of 0.15 mg/kg of Dexamethasone intravenously with a maximum dose of 5 mg
  Interventions: Drug: Dexamethasone
- Sodium chloride (Placebo Comparator): Single intraoperative administration of Sodium Chloride (NaCl) 0.9% intravenously
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Dexamethasone — Is usually commercialized as dexamethasone phosphate as solution for injection
  Arms: Dexamethasone
Drug: Sodium chloride — prepared in the same intravenous volume to mimic experimental arm
  Arms: Sodium chloride

SUMMARY:
Tonsillectomy is one of the most frequently performed surgical interventions in children. However, it is associated with a high incidence of PostOperative Nausea and Vomiting (PONV), severe pain and haemorrhage.

There is strong evidence on the efficacy of Dexamethasone in reducing the incidence of PONV and pain after tonsillectomy, which led to consider this drug as a first line treatment in routine anaesthesia practice in such surgical setting. However, in the last decade, there have been arguments about the potential role of Dexamethasone in increasing the risk of postoperative bleeding in children and studies addressing the haemorrhage risk following administration of Dexamethasone for tonsillectomy are inconclusive.Thus, this study is aimed at providing evidence for the safety profile of Dexamethasone with regard to the risk of post-tonsillectomy bleeding in children when administered as a single intraoperative dose.

DETAILED DESCRIPTION:
This double-blind (investigator-surgeon-patient blinded), randomized, placebo control, multicentre, international, pragmatic, non-inferiority trial is designed to to provide evidence of the Dexamethasone safety profile with regard to the risk of post-tonsillectomy bleeding in children when administered as a single intraoperative dose of 0.15mg/kg. The study is also aimed at characterizing whether the co-administration of non steroidal anti-inflammatory drugs for analgesia potentiates the risk of postoperative haemorrhage.

Sample size estimation is based on the definition of a minimal clinically important difference between the 2 groups of treatment (dexamethasone or normal saline) to be equal to 2% (non-inferiority margin). Thus, 3'794 children in total will be included with 1'897 children in each treatment group.

The follow-up will be performed by the parents via an "Application" for Android and Apple that has been developed specifically for this study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 2 to 13 years admitted for tonsillectomy/ tonsillotomy with or without adenoidectomy
* Parents or legal responsible person willing and capable to follow data collection by the application (Android and iPhone) developed for this study

Exclusion Criteria:

* Children under Aspirin or any other anticoagulants with or without Congenital Heart Disease
* Children with any bleeding disorders (ex. Haemophilia, Von Willebrand Disease)

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 523 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Reoperation for postoperative bleeding | Up to 30 days
  bleeding requiring surgical revision

SECONDARY OUTCOMES:
Respiratory complications | Intraoperative and up to 2 hours postoperative
  7) Incidence of perioperative respiratory critical events: laryngospasm, bronchospasm, stridor, bronchial aspiration, hypoxia (Saturation in oxygen<90% for 2 minutes)
Pain scores | Up to 7 days after surgery
  Assessment of pain scores at the hospital with the total score for the FLACC (Face, Legs, Activity, Cry, Consolability) scale for children less than 2 years of age and by the numeric pain rating scale above. Then at home, assessment by parents with the short version of the parents postoperative pain measurement.
Postoperative nausea, vomiting and retching | 3 intervals: 0-2 hours, 2-6 hours and 6-24 hours postoperatively
  2) Number of postoperative nausea and vomiting (PONV) and retching: during the stay at hospital with a maximum of 24 hours post-extubation
Morbidity | Up to 30 days
  Any admission to high dependency unit or ICU, readmission for following reasons: Ear, Nose and Throat infection, dehydration, pulmonary infection, other pulmonary complications, seizure or bleeding not requiring reoperation

CONTACTS AND LOCATIONS:
Locations (2):
- Queen Elizabeth Hospital of Montreal, Mc Gill, Montreal, Quebec, Canada
- geneva Children's Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Up to 2 years following study completion
Access Criteria: Data access requests from National coordinators or from local investigators will be examined by the steering committee and an agreement will be signed prior to Data access